CLINICAL TRIAL: NCT04344821
Title: Effects of Repeated Short-Term Diets on Weight Loss in Women Participating in the Curves Fitness Program
Brief Title: Curves 30/30 Study
Acronym: C-30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: Curves International (Industry)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB2008-0480
Record Dates: First submitted 2020-04-09; First posted 2020-04-14 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled, repeated measures intervention trial
Who Masked: Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Placebo Comparator): No diet or exercise intervention
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Placebo
- No Diet plus Exercise (Experimental): No diet, exercise only intervention
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Placebo
- High Protein Diet plus Exercise (Experimental): High protein diet and exercise intervention
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Placebo
- High Carbohydrate Diet plus Exercise (Experimental): High carbohydrate diet and exercise intervention
  Interventions: Dietary Supplement: Curves Calcium; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Curves Calcium — Dietary Supplement: Curves Calcium
  Curves Essential Bio-Available Calcium (providing 800 mg/d of calcium [as calcium citrate malate and calcium citrate], 400 IU of Vitamin D, 300 mg/d of magnesium, 4 mg/d of zinc, 2 mg/d of copper, 2 mg/d of manganese, 198 mg/d of potassium, 100 mg/d of trace mineral complex, and 2 mg/d of boron)
Dietary Supplement: Placebo — Dextrose Placebo

SUMMARY:
The purpose of this study is to determine whether following a high carbohydrate/low fat diet or high protein/low fat diet for 30-days several times during six months of participating in the Curves fitness and diet program with or without dietary calcium supplementation promotes stepwise reductions in body weight, improvements in body composition, and/or improvements in markers of fitness and health.

DETAILED DESCRIPTION:
The Curves International fitness and weight loss program has become a very popular means of promoting health and fitness among women. The program involves a 30-minute circuit training program and a weight management program involving periods of moderate caloric restriction (1,200 to 1,600 calories per day) followed by short periods of higher caloric intake (2,600 calories per day). The program is designed to promote a gradual reduction in body fat while increasing strength and muscle mass/tone. Researchers in the Exercise & Sport Nutrition Laboratory (ESNL) at Texas A&M University have conducted an extensive study on the effectiveness and safety of the Curves fitness and diet program. Results of this initial study have shown that the program promotes weight loss, improves markers of health, and improves fitness. However, we feel that the program may be even more effective with some additional nutritional interventions. Calcium has been shown to slow bone loss and more recently has been found to help promote fat loss. If this is the case, supplementing the diet with calcium may promote greater benefits in women participating in the Curves fitness and diet program. The purpose of this study is to determine whether following a high carbohydrate/low fat diet or high protein/low fat diet for 30-days several times during six months of participating in the Curves fitness and diet program with or without dietary calcium supplementation promotes stepwise reductions in body weight, improvements in body composition, and/or improvements in markers of fitness and health.

ELIGIBILITY:
Inclusion Criteria:

* Participant is female;
* Participant is post-menopausal;
* Participant is between the ages of 18 and 45;
* Participant is sedentary, overweight (BMI > 27) and post-menopausal;

Exclusion Criteria:

* Participant has any metabolic disorders including known electrolyte abnormalities, heart disease, arrhythmias, diabetes, or thyroid disease;
* Participant has a history of hypertension, hepatorenal, musculoskeletal, autoimmune or neurological disease;
* Participant is taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive or androgenic medications;
* Participant has taken ergogenic levels of nutritional supplements that may affect muscle mass (i.e., creatine, HMB, etc.), anabolic/catabolic hormone levels (i.e., androstenedione, DHEA, etc.) or weight loss (i.e., ephedra, thermogenics, etc.) within three months prior to the start of the study;
* Participant is consistently taking 500 mg or more of a Calcium supplement per day;
* Participant is receiving Hormone Replacement Therapy (HRT);
* Participant is involved in a planned exercise program within 3 - 6 months prior to the start of the study;
* Participant has lost > 20 lbs. within the last 3 - 6 months;

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Sedentary and overweight female participants between the ages of 18 and 45 participated in this study.
Enrollment: 57 (Actual)
Dates: Start 2009-05-18; Primary Completion 2012-05-03 (Actual); Study Completion 2012-05-03 (Actual)

PRIMARY OUTCOMES:
Body Composition: Body Fat | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (% body fat) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Fat Free Mass | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (fat free mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Bone Mass | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (bone mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Fat Mass | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (fat mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Lean Mass | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (lean mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Body Weight | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in body composition (body weight) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)

SECONDARY OUTCOMES:
Energy Homeostasis: Resting Energy Expenditure (REE) | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in REE obtained via metabolic cart and expressed in absolute (kcal/d) and relative terms kcals/kg/d) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Energy Homeostasis: Respiratory Exchange Ratio (RER) | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in RER as an indicator of carbohydrate and fat oxidation analyzed with related resting energy expenditure outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Strength: 1 Repetition Maximum (1 RM) Bench Press | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in bench press 1 RM obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Strength: 1 Repetition Maximum (1 RM) Leg Press | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in bench press 1 RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1 RM) Bench Press Endurance Test | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in total repetitions at 80% of 1 RM obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1 RM) Leg Press Endurance Test | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in total repetitions at 80% of 1 RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Cardiac Variable: Resting Electrocardiogram (ECG) | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in resting ECG obtained via electrodes and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Cardiac Variable: Graded Exercise Test (GXT) | Measured prior to supplementation (Pre), and after 3, and 6 months
  Changes in exercise capacity obtained via a treadmill test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Heart Rate (RHR) | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in resting heart rae (RHR) obtained via a blood pressure meter and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Systolic Blood Pressure (SBP) | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in resting systolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Diastolic Blood Pressure (DBP) | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in resting diastolic blood pressure (mmHg) analyzed with related resting hemodynamic outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist Circumference | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in waist circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Hip Circumference | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in hip circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist to Hip Ratio | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in the ratio of waist to hip (waist/hip circumference) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Fasting Glucose | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in glucose obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Cholesterol | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: HDL Cholesterol | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in HDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Cholesterol to HDL Ratio | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in cholesterol to HDL ratio obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: LDL Cholesterol | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in LDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Triglycerides | Measured prior to supplementation (Pre), and after 1, 2, 3, 4, 5 and 6 months
  Changes in triglycerides obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise & Sport Nutrition Laboratory, College Station, Texas, United States

IPD SHARING:
Plan to Share IPD: No